CLINICAL TRIAL: NCT02059603
Title: A Randomized Clinical Trial of Electroacupuncture Versus Fast-track Perioperative Program for Reducing Duration of Postoperative Ileus and Hospital Stay After Laparoscopic Colorectal Surgery
Brief Title: Electroacupuncture Versus Fast-track Perioperative Program for Laparoscopic Colorectal Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Simon S. M. Ng, Professor of Surgery, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2013.009
Record Dates: First submitted 2014-02-10; First posted 2014-02-11 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Postoperative Ileus
Keywords: Electroacupuncture; Fast track program; Postoperative ileus; Laparoscopic surgery; Colorectal surgery; Randomized controlled trial; Hospital stay
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electroacupuncture (Experimental): Bilateral acupoints relevant to the treatment of abdominal pain, abdominal distension, and constipation, including Zusanli (stomach meridian ST-36), Sanyinjiao (spleen meridian SP-6), Hegu (large intestine meridian LI-4), and Zhigou (triple energizer meridian TE-6), will be used. Electric stimulation at a frequency of 50 Hz will be employed to the acupuncture needles.
  Interventions: Procedure: Electroacupuncture
- Fast-track program (Active Comparator): The design of this program is based on the consensus between our surgeons, anesthetists, physiotherapists, dietitians, and nurses, who have reviewed the relevant literature and made appropriate adjustments to suit the local situation.
  Interventions: Procedure: Fast-track program

INTERVENTIONS:
Procedure: Electroacupuncture
  Arms: Electroacupuncture
Procedure: Fast-track program
  Arms: Fast-track program

SUMMARY:
Background: Our previous study demonstrated that electroacupuncture at Zusanli, Sanyinjiao, Hegu, and Zhigou reduces the duration of postoperative ileus and hospital stay after laparoscopic colorectal surgery within a traditional perioperative care setting. Recent evidence also suggested that a 'fast-track' perioperative program may help accelerate recovery after colorectal surgery. As electroacupuncture is simpler to implement and less labor intensive, it may be the preferred adjunct therapy if it is proven to be noninferior to fast-track program in reducing the duration of postoperative ileus and hospital stay after laparoscopic colorectal surgery.

Objectives: To compare the efficacy of electroacupuncture and fast-track program in reducing the duration of postoperative ileus and hospital stay after laparoscopic colorectal surgery.

Design: Prospective, randomized, noninferiority trial.

Subjects: One hundred sixty-four consecutive patients undergoing elective laparoscopic resection of colonic and upper rectal cancer will be recruited.

Interventions: Patients will be randomly allocated to receive either: (A) electroacupuncture with traditional perioperative care; or (B) fast-track program without acupuncture.

Outcome measures: Primary outcome: time to defecation. Secondary outcomes: duration of hospital stay, time of first passing flatus, time to resume diet, pain scores, analgesic requirement, morbidity, and medical costs.

Conclusions: This study will determine if electroacupuncture is noninferior to fast-track program in reducing the duration of postoperative ileus and hospital stay after laparoscopic colorectal surgery. Electroacupuncture may be the preferred perioperative adjunct therapy to laparoscopic colorectal surgery because it is simpler to implement and less labor intensive than fast-track program.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients undergoing elective laparoscopic resection of colonic and upper rectal cancer
* Age of patients between 18 and 80 years
* Patients with American Society of Anesthesiologists (ASA) grading I-II
* Patients with no severe physical disability
* Patients who require no assistance with the activities of daily living
* Informed consent available

Exclusion Criteria:

* Patients undergoing laparoscopic low anterior resection with total mesorectal excision, abdominoperineal resection, or total/proctocolectomy
* Patients with planned stoma creation
* Patients undergoing emergency surgery
* Patients with evidence of peritoneal carcinomatosis
* Patients with previous history of midline laparotomy
* Patients who are expected to receive epidural opioids for postoperative pain management
* Patients with cardiac pacemaker
* Patients who are allergic to the acupuncture needles

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Time to defecation | Up to 1 month
  Measured in hours, from the time the laparoscopic surgery ends till the first observed passage of stool.

SECONDARY OUTCOMES:
Total postoperative hospital stay | Up to 1 month
  Including hospital stay of patients who are readmitted within 30 days after surgery.
Time of first passing flatus reported by the patients | Up to 1 month
Time that the patients tolerated solid diet | Up to 1 month
Time to walk independently | Up to 1 month
Pain scores on visual analog scale | Up to 1 month
  From 0 which implies no pain at all, to 100 which implies the worst pain imaginable; assessed at 4, 12, 24, 48, and 72 hours after surgery.
Morbidity | Up to 1 month
Mortality | Up to 1 month
Readmission rate | Up to 1 month
Quality of life | Up to 1 month
  Quality of life at 2 and 4 weeks after surgery, measured by SF-36, EORTC QLQ-C30 and QLQ-CR38 questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Simon S. M. Ng, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, China